CLINICAL TRIAL: NCT06504017
Title: FUS-TB VS COG-TB in Prostate Cancer With PI-RADS 4 Small Lesions - a Predictive, Multi-center, Exploring Study
Brief Title: FUS-TB VS COG-TB in Small Lesions of Prostate Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Huai'an First People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024-SR-359
Record Dates: First submitted 2024-07-10; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COG-TB: Cognitive Fusion guided prostate targeted Biopsy (Other): Targeted Biopsy 4 cores under cognitive fusion ultrasound
  Interventions: Procedure: COG-TB: Cognitive Fusion guided prostate targeted Biopsy
- FUS-TB: MRI-TRUS Fusion guided prostate targeted Biopsy (Experimental): Targeted Biopsy 4 cores under MRI-TRUS Fusion ultrasound
  Interventions: Procedure: FUS-TB: MRI-TRUS Fusion guided prostate targeted Biopsy

INTERVENTIONS:
Procedure: COG-TB: Cognitive Fusion guided prostate targeted Biopsy — Cognitive Fusion guided targeted Biopsy 4 cores under cognitive fusion ultrasound
  Arms: COG-TB: Cognitive Fusion guided prostate targeted Biopsy
Procedure: FUS-TB: MRI-TRUS Fusion guided prostate targeted Biopsy — MRI-TRUS Fusion guided targeted Biopsy 4 cores under cognitive fusion ultrasound
  Arms: FUS-TB: MRI-TRUS Fusion guided prostate targeted Biopsy

SUMMARY:
To compare the positive detection rates of COG-TB vs FUS-TB for prostate cancer with PI-RADS 4 small lesions.

DETAILED DESCRIPTION:
Prostate cancer (PCA) is the most frequent malignancy in male urogenital system. According to the World Health Organization's 2020 GLOBOCAN statistics, there are approximately 1.4 million new cases and 375,000 deaths worldwide. PCa is the second most common tumor in male patients after lung cancer and ranks fifth among cancer causes of death.

Currently, prostate specific antigen ( PSA ), digital rectal examination (DRE), multi-parametric magnetic resonance imaging (mpMRI), prostate specific membrane antigen positron emission Tomography/computed tomography (PSMA PET/CT) and other detection methods have played an important role in the diagnosis of PCa, but the gold standard for confirming PCa is the histopathological examination of prostate biopsy. Performing mpMRI before biopsy can help detect and locate prostate cancer with ISUP grade ≥2. Studies have shown that the prostate imaging reporting and data system (PI-RADS) may help improve the detection of clinically significant cancers. Biopsy should be considered when PI-RADS score 4 or 5.

This clinical study intends to use the mpMRI-TRUS image fusion ultrasound system to assist in guiding FUS-TB, comparing to COG-TB to evaluate the application value of mpMR-TRUS image fusion in the detection of PCa in prostate biopsy.

ELIGIBILITY:
Inclusion Criteria:

* 1) male who are between 18 to 80 years old; 2) meet any of the following criteria:

  1. suspicious nodules of prostate under digital rectal examination(DRE), with any PSA value;
  2. PSA≥10μg/L;
  3. 4μg/L≤PSA<10μg/L,f/t PSA≤0.16; 3) suspicious lesions under mpMRI, at least one lesion <5mm, PI-RADS 4; 4) good compliance; 5) must sign the informed consent form.

Exclusion Criteria:

* 1) diagnosed prostate cancer or acute prostatitis; 2) acute infection, or clinically significant urinary tract infection; 3) performed prostate puncture within 1 month; 4) cardiac insufficiency; 5) having high risk of bleeding or taking anticoagulants for a long time; 6) severe internal or external hemorrhoids, perianal or rectal lesions; 7) having severe osteoarticular diseases that can not be performed lithotomy; 8) hypertensive crisis; 9) patients who should not be anesthetized; 10) patients with mental illness or mental disorders and unable to understand the informed consent; 11) patients with electronic devices such as built-in artificial pacemaker, cochlear implants or nerve stimulators; 12) other surgical contraindications, or those considered unsuitable by the investigators.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The prostate is unique to men
Enrollment: 200 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
detection rate of any PCa | 1 week (after pathology）
  detection rate of any prostate cancer

SECONDARY OUTCOMES:
detection rate(cs PCa and PCa) of TBx | 1 week (after pathology）
  detection rate for PI-RADS 4 small lesion (<5mm) under MRI-TRUS fusion

CONTACTS AND LOCATIONS:
Overall Officials: Shangqian Wang, PhD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University

IPD SHARING:
Plan to Share IPD: No